CLINICAL TRIAL: NCT00389688
Title: Randomized Phase II Study of Pemetrexed and Cisplatin as Either Induction or Adjuvant Chemotherapy in Stage IB-II Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Pemetrexed Disodium and Cisplatin Before or After Surgery in Treating Patients With Stage IB or Stage II Non-Small Cell Lung Cancer That Can be Removed by Surgery
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: low accrual
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: EORTC-08051; EORTC-08051; 2005-003822-25 (EudraCT Number)
Record Dates: First submitted 2006-10-18; First posted 2006-10-19 (Estimated); Last update posted 2012-07-18 (Estimated); Status verified 2012-07

CONDITIONS: Lung Cancer
Keywords: stage I non-small cell lung cancer; stage II non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Cisplatin; Pemetrexed; Chemotherapy, Adjuvant; Neoadjuvant Therapy

INTERVENTIONS:
Drug: cisplatin
Drug: pemetrexed disodium
Procedure: adjuvant therapy
Procedure: conventional surgery
Procedure: neoadjuvant therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as pemetrexed disodium and cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed. Giving combination chemotherapy after surgery may kill any tumor cells that remain after surgery. It is not yet known whether combination chemotherapy is more effective before or after surgery in treating non-small cell lung cancer.

PURPOSE: This randomized phase II trial is studying the side effects of pemetrexed disodium and cisplatin and comparing how well they work when given before or after surgery in treating patients with stage IB or stage II non-small cell lung cancer that can be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the tolerability (in terms of drug delivery and toxicity) of neoadjuvant vs adjuvant chemotherapy comprising cisplatin and pemetrexed disodium in patients with resectable stage IB or II non-small cell lung cancer.

Secondary

* Determine the overall toxicity of this regimen in these patients.
* Determine the progression-free and overall survival of patients treated with this regimen.
* Determine the overall clinical response rate, pathologic complete response, and resectability rate in patients treated with neoadjuvant chemotherapy.
* Determine the surgical morbidity and mortality of patients treated with these regimens.
* Determine the fraction of patients in the adjuvant arm that receives chemotherapy.

OUTLINE: This is a randomized, open-label, multicenter study. Patients are stratified according to institution, histological subtype (squamous vs nonsquamous) and clinical stage (IB vs II). Patients are randomized to 1 of 2 treatment arms.

* Arm I (neoadjuvant chemotherapy): Patients receive cisplatin IV over 3-6 hours and pemetrexed disodium IV on day 1. Treatment repeats every 21 days for up to 3 courses in the absence of disease progression or unacceptable toxicity. Four to six weeks after completion of chemotherapy, patients undergo surgery.
* Arm II (adjuvant chemotherapy): Patients undergo surgery. Beginning 4-8 weeks after surgery, patients receive cisplatin and pemetrexed disodium as in arm I.

After completion of study treatment, patients are followed periodically for 5 years and then annually thereafter.

PROJECTED ACCRUAL: A total of 132 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Pathologically confirmed non-small cell lung cancer (NSCLC)

  * Stage IB or II disease
* Resectable disease
* At least 1 measurable lesion
* No mediastinal involvement by mediastinoscopy and/or positron emission tomography with fludeoxyglucose F 18 scan
* No evidence of metastatic disease

PATIENT CHARACTERISTICS:

* WHO performance status 0-2
* Absolute neutrophil count > 1,500/mm³
* Platelet count > 100,000/mm³
* Hemoglobin > 10 g/dL
* Creatinine clearance ≥ 60 mL/min
* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* Alkaline phosphatase ≤ 3.0 times ULN
* AST and ALT ≤ 3.0 times ULN
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No other malignant disease, except for the following:

  * Basocellular carcinoma of the skin
  * Adequately treated carcinoma in situ of the cervix
  * Low-grade prostate cancer
  * Other cancer for which the patient has been disease-free for ≥ 5 years
* No congestive heart failure or angina pectoris unless medically controlled
* No myocardial infarction within the past 6 months
* No uncontrolled hypertension or arrhythmia
* No active uncontrolled infection requiring antibiotics
* No illness or medical condition that would preclude study participation
* No pre-existing motor or sensory neurotoxicity ≥ grade 2

PRIOR CONCURRENT THERAPY:

* No prior surgery for NSCLC
* No prior or other concurrent chemotherapy for NSCLC
* No prior or concurrent radiotherapy for NSCLC
* No concurrent immunotherapy
* No concurrent targeted agents
* No concurrent hormonal cancer therapy
* No concurrent routine colony-stimulating factor (e.g., prophylactic filgrastim [G-CSF])
* No aspirin or nonsteroidal anti-inflammatory drugs within 5 days before or after chemotherapy
* No other concurrent experimental treatments
* No other concurrent anticancer treatments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2006-08; Primary Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Successful treatment delivery
Toxicity (no grade 4) during chemotherapy

SECONDARY OUTCOMES:
Overall toxicity (all grades)
Progression-free survival and overall survival
Overall clinical response rate (neoadjuvant chemotherapy arm)
Pathologic complete response (neoadjuvant chemotherapy arm)
Resectability rate (neoadjuvant chemotherapy arm)
Surgical morbidity and mortality
Fraction of patients that actually receives chemotherapy (adjuvant chemotherapy arm)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Germonpre, MD, Study Chair — University Hospital, Antwerp
Locations (1):
- Universitair Ziekenhuis Antwerpen, Edegem, Belgium